CLINICAL TRIAL: NCT05395026
Title: Systematic Evaluation of Vagus Nerve Stimulation Parameters on Cardiac Rhythm, Laryngeal Muscle Electromyography, and Vagus Nerve Activation in Acute and Chronic Implantations
Brief Title: Systematic Evaluation of VNS Parameters
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: current funding ended
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00103473
Record Dates: First submitted 2022-05-18; First posted 2022-05-27 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational Stimulation Parameters (Experimental)
  Interventions: Other: electrical stimulation of vagus nerve

INTERVENTIONS:
Other: electrical stimulation of vagus nerve — VNS electrical stimulation parameters (pulse duration, pulse amplitude, and pulse frequency) will be systematically changed to determine the effect on vagus nerve activation, laryngeal muscle contraction, and heart rate.

SUMMARY:
The goal of this study is to measure the activation of the vagus nerve and the side effects of vagus nerve stimulation (VNS) (neck muscle contractions, changes in heart rate) across a range of stimulation parameters typically used in VNS therapy for epilepsy (pulse durations, pulse amplitudes, pulse repetition rates). This mapping of the parameter space may inform future device programming to improve electrical activation of the vagus nerve and/or to reduce side effects, and it may be used for validation of computational models. The study will recruit adult participants with epilepsy who are undergoing surgery either for an initial implant of a VNS device or for replacement of the implanted pulse generator (IPG) due to battery depletion. During surgery, the study will involve stimulating the vagus nerve via the standard implanted clinical VNS electrodes over a range of stimulation parameters while recording the activity of the vagus nerve (electroneurogram (ENG)), electromyogram (EMG) response of neck/throat muscles, and the heart rate (electrocardiogram (EKG)). Stimulation parameters will be within the ranges used for clinical therapy and below limits established for non-damaging electrical stimulation.

DETAILED DESCRIPTION:
This study will recruit adult participants with epilepsy who are undergoing planned surgery either for an initial implant of a vagus nerve stimulation (VNS) device or for replacement of their VNS implanted pulse generator (IPG) due to battery depletion. The primary study goals are to measure the activation of the vagus nerve and the side effects of vagus nerve stimulation (neck muscle contractions, changes in heart rate) across a range of stimulation parameters typically used in VNS therapy for epilepsy. This mapping of the parameter space may inform future device programming to improve electrical activation of the vagus nerve and/or to reduce side effects. All study participants will be assigned to a single study group and will complete the same study procedures.

The research study will take place during VNS surgery. For participants undergoing a first VNS implant surgery, once the vagus nerve is exposed and before placing the VNS electrodes, the investigators may image the nerve with ultrasound. Mapping of the parameter space will then occur after placement of the cuff electrodes around the cervical vagus nerve for participants undergoing a first VNS implant surgery or removal of the IPG with the depleted battery for patients undergoing IPG replacement surgery. Temporary sterile extension wires will connect the implanted VNS electrode to the research stimulation system. Research procedures will involve stimulating the vagus nerve through the standard implanted clinical VNS electrodes over a range of stimulation parameters. At the same time, the investigators will record how changes in stimulation affect the activity of the vagus nerve (measured by electroneurogram (ENG)), the response of the neck and throat muscles (by electromyogram (EMG)) and the heart rate (by electrocardiogram (EKG)). Several stimulation trials will be conducted with different VNS parameters (pulse duration, pulse amplitude, and pulse repetition rate) delivered in randomized order. Stimulation parameters will be within the ranges used for clinical therapy and will not exceed those that produce a 25% reduction in heart rate. Measurements will be made during 10 to 60 second trials, in which stimulation will be off for the first section (baseline), on for the second section (responses to stimulation), and off for the final section (recovery). The stimulus waveform will be a charge-balanced biphasic pulse, with values of charge density (D) limited to values below the nondamaging limits that are well-established in literature.

ELIGIBILITY:
Inclusion Criteria:

* adult epilepsy patients undergoing VNS electrode implantation or implanted pulse generator (IPG) replacement surgery
* in good health
* neurologically stable aside from epilepsy
* able to provide informed consent

Exclusion Criteria:

* patients with another implanted electrical device (besides VNS)
* a history of heart conditions that the surgeon considers a contraindication to study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
stimulation amplitude threshold | During procedure (30 minutes)
  The stimulation amplitude threshold is the amplitude when vagus nerve stimulation (VNS) activates the laryngeal muscles and has potential to cause subject discomfort during stimulation. The stimulation amplitude threshold will be measured with the NIM-EMG endotracheal tube recording, and the threshold will be determined as the amplitude that causes the first evoked potential in the laryngeal muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Warren M Grill, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cogan SF, Ludwig KA, Welle CG, Takmakov P. Tissue damage thresholds during therapeutic electrical stimulation. J Neural Eng. 2016 Apr;13(2):021001. doi: 10.1088/1741-2560/13/2/021001. Epub 2016 Jan 20. PMID 26792176
- [Background] Kumsa D, Steinke GK, Molnar GF, Hudak EM, Montague FW, Kelley SC, Untereker DF, Shi A, Hahn BP, Condit C, Lee H, Bardot D, Centeno JA, Krauthamer V, Takmakov PA. Public Regulatory Databases as a Source of Insight for Neuromodulation Devices Stimulation Parameters. Neuromodulation. 2018 Feb;21(2):117-125. doi: 10.1111/ner.12641. Epub 2017 Aug 7. PMID 28782181